CLINICAL TRIAL: NCT00676637
Title: A Pilot Study of Adherence Assessment With the Travalert™ Dosing Aid in Patients With Ocular Hypertension or Primary Open-Angle Glaucoma Who Are Treated With the Travoprost/Timolol Maleate Fixed Combination Every Evening
Brief Title: Glaucoma Adherence Study
Acronym: GAS
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: EMD-07-01; EMD-07-02 (Other: Alcon)
Record Dates: First submitted 2008-05-12; First posted 2008-05-13 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Ocular Hypertension; Primary Open Angle Glaucoma
Keywords: Adherence; Compliance; Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle; Patient Compliance; Glaucoma | interventions — Travoprost; Timolol; Duotrav

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Travalert with DuoTrav: One drop in study eye(s) once daily in the evening for four months
  Interventions: Drug: Travoprost 0.004%/timolol 0.05% fixed combination eye drops (DuoTrav); Device: Travalert Dosing Aid

INTERVENTIONS:
Drug: Travoprost 0.004%/timolol 0.05% fixed combination eye drops (DuoTrav) — One drop in study eye(s) once daily in the evening for four months
  Other Names: DuoTrav
Device: Travalert Dosing Aid — Approved device used with DuoTrav and intended to provide an objective system for quantifying dosing and improving patient adherence

SUMMARY:
The purpose of this study is evaluate adherence to DuoTrav® when reinforced by the use of the Travalert™ Dosing Aid.

DETAILED DESCRIPTION:
This study was conducted in France, UK, Italy, and Netherlands. An identical study was conducted in Spain under Protocol ID EMD-07-02. A combined enrollment number is presented.

ELIGIBILITY:
Inclusion:

* Provide informed consent.
* Able to follow instructions and be willing and able to attend required study visits.
* Able to read and complete study questionnaires.
* Clinical diagnosis of ocular hypertension, or primary open-angle, pigment dispersion or exfoliation glaucoma in at least one eye.
* Intraocular pressure considered safe, in both eyes, assuring clinical stability of vision and the optic nerve throughout the trial.
* Currently treated with DuoTrav alone, dosed in the evening for at least for 30 days, at Visit 1.
* Best corrected visual acuity of 20/200 Snellen or better in each eye.
* Intraocular pressure ≤ 30 mm Hg in both eyes.
* Evidence causing the investigator to consider the patient to be non-adherent, at some level, to their glaucoma medication.
* Agree that their adherence could be improved by the intervention with the dosing aid described in this study.
* Other protocol-defined inclusion criteria may apply.

Exclusion:

* Presence of other primary or secondary glaucoma not listed in inclusion criterion.
* Any abnormality preventing reliable applanation tonometry in the study eye(s).
* Any known opacity or patient uncooperativeness that restricts adequate examination of the ocular fundus or anterior chamber of the study eye(s).
* Concurrent infectious/noninfectious conjunctivitis, keratitis or uveitis in either eye.
* Intraocular conventional surgery or laser surgery in study eye(s) less than three months prior to Visit 1.
* Risk of visual field or visual acuity worsening as a consequence of participation in the trial, in the investigator's best judgment.
* Progressive retinal or optic nerve disease from any cause.
* Women of childbearing potential not using reliable means of birth control.
* Women who are pregnant or lactating.
* A condition, which in the opinion of the Principal Investigator, would interfere with optimal participation in the study, or which would present a special risk to the patient.
* Participation in any other investigational study within 30 days prior to Visit 1.
* Known medical history of allergy, sensitivity or poor tolerance to any components of the preparations to be used in this trial that is deemed clinically significant in the opinion of the Principal Investigator.
* Unwillingness to risk the possibility of darkened irides, eyelash changes or periocular pigmentation.
* History of, or at risk for uveitis or cystoid macular edema (CME).
* Any physical disability which prevents the accurate use of the Travalert™ dosing aid.
* Unable to accurately instill the travoprost/timolol fixed combination in the evening.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were selected from five study sites in the European Union.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2008-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in Intraocular Pressure at 4 months | Baseline, 4 months
  As measured by Goldmann applanation tonometry

CONTACTS AND LOCATIONS:
Overall Officials: Anna Grau, Study Director — Alcon Research
Locations (4):
- France, Paris, France
- Milan, Milan, Italy
- Maastricht, Maastricht, Netherlands
- London, London, United Kingdom